CLINICAL TRIAL: NCT00782405
Title: Effect of Quetiapine XR on Sleep in Patients With Major Depression, as Compared With Mirtazapine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Technical University of Munich, TechnischeUM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D114432C00027
Record Dates: First submitted 2008-10-24; First posted 2008-10-31 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Sleep
Keywords: antidepressant action; clinical psychopharmacology
MeSH Terms: interventions — Quetiapine Fumarate; Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): quetiapine
  Interventions: Drug: quetiapine
- 2 (Active Comparator): mirtazapine
  Interventions: Drug: mirtazapine

INTERVENTIONS:
Drug: quetiapine — XR, 150-300mg
  Arms: 1
Drug: mirtazapine — 30-45 mg
  Arms: 2

SUMMARY:
The purpose of this study is to examine the effects of (a) quetiapine XR and (b) mirtazapine on sleep when given as an antidepressant (monotherapy). We hypothesize that (a) quetiapine XR has an immediate and lasting positive effect on sleep in depressed patients which does not differ from the impact of mirtazapine on sleep in this group of patients; (b) in the context of a secondary objective, we expect an antidepressant effect of quetiapine XR which is equivalent to that of mirtazapine.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. A diagnosis of Major depressive disorder by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, revised (DSM-IV-R)
3. Clinically significant sleep disturbance (PSQI total score > 5)
4. Females and males aged 18 to 65 years
5. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrolment
6. Able to understand and comply with the requirements of the study
7. Minimum score in the HAMD-21 scale: 18

Exclusion Criteria:

1. Pregnancy or lactation
2. Any DSM-IV-R Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate and / or mirtazapine, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampicin, St. John's Wort, and glucocorticoids
7. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
8. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV-R criteria
9. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV-R criteria within 4 weeks prior to enrolment
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
12. Involvement in the planning and conduct of the study
13. Previous enrolment or randomisation of treatment in the present study.
14. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
15. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
16. An absolute neutrophil count (ANC) of ≤ 1.5 x 109 per liter
17. Respiratory distress index during the 1st polysomnography > 10
18. Periodic leg movement / arousal index during the 1st polysomnography > 10

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
sleep effiency

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Wiegand, Prof., Principal Investigator — Sleep Disorders Center
Locations (1):
- Sleep Disorders Center, Munich, Bavaria, Germany